## NCT03232801

Title: A Mindfulness-based Intervention for Older Women with Low Sexual Desire

Date: August 1, 2022

Statistical analysis:

We assessed satisfaction and likelihood of recommending the group to another woman with low libido at 7 weeks (primary outcome). We assessed sexual function [Female Sexual Function Index (FSFI)] and sexual distress [Female Sexual Distress Scale-Revised (FSDS-R)] at 12 weeks (exploratory outcomes). We used chi squared statistics to examine differences in primary outcomes between groups. We constructed linear regression models to compare changes in FSFI and FSDS-R from baseline to 12 weeks for each group.